CLINICAL TRIAL: NCT05974514
Title: Investigation of Physical Parameters Influencing Body Awareness in Adults With Obesity: An Observational, Controlled Study
Brief Title: Body Awareness in Adults With Obesity
Status: Completed | Type: Observational
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Çağdaş IŞIKLAR, Lecturer, MSc Physiotherapist (PT), Fenerbahce University
Other Study IDs: 29.12.2022/141
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Obesity
Keywords: Obesity; Body awareness; Physical activity; Balance; Proprioception; Reaction time
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to examine the level of body awareness in individuals with obesity and investigate the parameters associated with body awareness. In addition, compare these parameters with healthy subjects with normal weight. The main questions it aims to answer are:

* How is body awareness affected compared to healthy individuals?
* Is physical activity level, dynamic balance, proprioception, and reaction time related to body awareness in individuals with obesity?
* Is there any difference between obese and normal-weight individuals in terms of physical activity level, dynamic balance, proprioception, and reaction time?

ELIGIBILITY:
Inclusion Criteria:

* Adults with obesity ((BMI) ≥ 30 kg/m2) aged 18-65 years, who did not receive obesity-related treatment 6 months before the study
* Healthy adults with normal weight (BMI: 18.5-24.9 kg/m2).

Exclusion Criteria:

* Musculoskeletal, neurological, and rheumatological disorders (fractures, sprains or strains, spine surgery, advanced respiratory or orthopaedic problems),
* Malignancy and pregnancy within the last 12 months, which might interfere with evaluations

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include 30 individuals with obesity and 30 healthy subjects. The individuals with obesity will be selected from internal medicine or dietitian clinics in Istanbul/Turkey.
  Healthy subjects will be age and sex-matched to serve as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Body Awareness | Baseline (Only 1 time)
  The Body Awareness Questionnaire will be used to assess body awareness. This questionnaire includes physical, emotional, and social aspects of a person's susceptibility to normal or abnormal bodily conditions and processes, questioning susceptibility to physical reactions. There are 18 statements in the questionnaire, each scored between 1 and 7 points (1=Not at all suitable for me, 7=Completely suitable for me). The total score is 126 and higher indicates a better body awareness level.

SECONDARY OUTCOMES:
Physical activity level | Baseline (Only 1 time)
  To evaluate self-reported physical activity level, International Physical Activity Questionnaire-Short Form (IPAQ-SF) will be used. The IPAQ-SF (7 questions) provides information about time spent on walking, moderate-intensity, and vigorous-intensity activities, as well as time spent sitting. The energy MET-minute score for these activities is calculated using standard MET values, which are as follows: Sitting: 1.5 MET, walking: 3.3 MET, moderate-intensity physical activity: 4.0 MET, vigorous-intensity physical activity: 8.0 MET.
  The total MET minutes per week are determined by taking the provided MET value and multiplying it by the total minutes spent engaging in the activity each day. Then, the MET minutes for all the days that the particular activity was performed are added up. Finally, the MET minutes from different activities are added up to get the total MET minutes per week. Physical activity level is categorized as low, moderate, and high.
Dynamic balance | Baseline (Only 1 time)
  Dynamic balance will be evaluated with the functional reach test. In this test, when standing upright, the distance covered by an extended arm during a complete forward reach, while ensuring a fixed supporting stance is measured.
Proprioception | Baseline (Only 1 time)
  The joint position sense assessment will be conducted using a Baseline bubble inclinometer to evaluate proprioception.
Reaction time | Baseline (Only 1 time)
  The Nelson Foot Reaction Test will be used to evaluate individuals' reaction speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Maltepe, Turkey (Türkiye)

REFERENCES:
- [Background] Karaca S, Bayar B. Turkish version of body awareness questionnaire: validity and reliability study. Türk Fizyoterapi ve Rehabilitasyon Dergisi. 2021;32(1):44-50.
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Healey EL, Allen KD, Bennell K, Bowden JL, Quicke JG, Smith R. Self-Report Measures of Physical Activity. Arthritis Care Res (Hoboken). 2020 Oct;72 Suppl 10(Suppl 10):717-730. doi: 10.1002/acr.24211. No abstract available. PMID 33091242
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Romero-Franco N, Montano-Munuera JA, Fernandez-Dominguez JC, Jimenez-Reyes P. Validity and Reliability of a Digital Inclinometer to Assess Knee Joint Position Sense in an Open Kinetic Chain. J Sport Rehabil. 2019 May 1;28(4):332-338. doi: 10.1123/jsr.2017-0221. Epub 2018 Dec 12. PMID 29252090
- [Background] Baert IAC, Lluch E, Struyf T, Peeters G, Van Oosterwijck S, Tuynman J, Rufai S, Struyf F. Inter- and intrarater reliability of two proprioception tests using clinical applicable measurement tools in subjects with and without knee osteoarthritis. Musculoskelet Sci Pract. 2018 Jun;35:105-109. doi: 10.1016/j.msksp.2017.11.011. Epub 2017 Nov 21. PMID 29174222
- [Background] Jung K, Kim Y, Chung Y, Hwang S. Weight-shift training improves trunk control, proprioception, and balance in patients with chronic hemiparetic stroke. Tohoku J Exp Med. 2014 Mar;232(3):195-9. doi: 10.1620/tjem.232.195. PMID 24646921
- [Background] Tamer K. Sporda fizyolojik fiziksel performansın ölçülmesi ve değerlendirilmesi. Ankara: Bağırgan Yayımevi; 2000